CLINICAL TRIAL: NCT03360019
Title: Accurate WiFi-Based Localization of Dementia Patients For Caregiver Support: Phase II
Brief Title: Accurate WiFi-Based Localization of Dementia Patients For Caregiver Support:
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Aster Labs, Inc (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB201702352 -N -A; OCR17448 (Other: OnCore); 5R44AG046944-03 (NIH)
Record Dates: First submitted 2017-11-27; First posted 2017-12-02 (Actual); Results first posted 2023-05-17 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Dementia, Vascular; Alzheimer Dementia; Lewy Body Dementia With Behavioral Disturbance
MeSH Terms: conditions — Dementia, Vascular; Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: Counterbalanced within-subject design. Specifically, each target patient will randomly be assigned to either have the technology or not have the technology applied for a period of three months, followed by three months of the opposite condition. Caregivers will provide caregiver ratings twice monthly during these two epochs.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Residents in memory care or skilled nursing Facility (Active Comparator)
  Interventions: Device: Activlink insole
- Resident in independent living setting (Active Comparator)
  Interventions: Device: Activlink insole
- Care Partners (Other)
  Interventions: Other: Activlink Phone Application

INTERVENTIONS:
Device: Activlink insole — Dementia patients will wear the provided insole inserted into their own shoes. The insole will have a small electronic sensor that measures acceleration, foot force, and/or orientation.
  Other Names: Location Monitoring Technology
  Arms: Resident in independent living setting; Residents in memory care or skilled nursing Facility
Other: Activlink Phone Application — Smartphone tool used for monitoring location
  Other Names: Location Monitoring Technology
  Arms: Care Partners

SUMMARY:
In this Phase II SBIR project we will enhance a wireless WiFi-based insole that was designed and successfully tested during a Phase I trial with elderly persons with dementia and their caregivers, and then investigate its efficacy in terms of caregiver activity, burden, and quality of life in Phase II. Evaluation will use semi-structured interviews and participant observation data collected from professional and family caregivers of patients with moderate or mild dementia.

DETAILED DESCRIPTION:
The efficacy of the Activlink system offering localization information to improve caregiver will be evaluated in two studies. Study 2a will use the insole system with dementia patients residing in skilled or memory care. Data regarding caregiving activity will be collected from their paid professional care providers. Study 2b will use participant localization data collected on 80 independently dwelling mild dementia patients. In this case data will be collected from their unpaid family caregivers. Both studies will result in evaluating the efficacy of the WiFi-based insole to provide caregivers with augmented patient awareness, helping to improve their immediate quality of life by reducing their direct burden of continuous oversight of their person in care.

ELIGIBILITY:
Inclusion Criteria:

Persons With Dementia Resides in memory care or skilled nursing

* Moderate dementia (MMSE of 10-18)
* Ambulatory (without or with cane, walker or wheelchair assist)
* A legal proxy that can provide consent

Persons With Dementia Resides in independent living setting in community.

* Mild dementia (MMSE of 19-25)
* Ambulatory (without or with cane, walker or wheelchair assist).
* Has a legal proxy that can provide consent.

Care Partners

* Speaks English
* Be 21 years of age or over
* Has at least three times per week direct contact with person with dementia (PWD)
* Consents to participate in the study

Exclusion Criteria:

* Is not fluent in written or spoken English
* Indicate an unwillingness to use the Activlink
* History of Major Mental Illness for patient or caregiver

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-01-27 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Smith, PhD, ABPP-cn, Principal Investigator — University of Florida
Locations (2):
- United States (2):
  - Oak Hammock Senior Living Center, Gainesville, Florida
  - Unversity of Florida, Gainesville, Florida

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Residents in Memory Care or Skilled Nursing Facility | Resident in Independent Living Setting | Care Partners
Started | 10 | 0 | 3
Completed | 2 | 0 | 3
Not Completed | 8 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0
Not completed — Pandemic caused suspension of study activities | 6 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Pandemic circumvented recruitment of independent living residents.
Groups:
- Total: Total of all reporting groups
Arm/Group | Residents in Memory Care or Skilled Nursing Facility | Resident in Independent Living Setting | Care Partners | Total
Number analyzed (Participants) | 10 | 0 | 3 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0 | 0
  Between 18 and 65 years | 1 |  | 3 | 4
  >=65 years | 9 |  | 0 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 |  | 3 | 10
  Male | 3 |  | 0 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 |  | 0 | 0
  Not Hispanic or Latino | 10 |  | 3 | 13
  Unknown or Not Reported | 0 |  | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0 | 0
  Asian | 0 |  | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0 | 0
  Black or African American | 0 |  | 0 | 0
  White | 10 |  | 3 | 13
  More than one race | 0 |  | 0 | 0
  Unknown or Not Reported | 0 |  | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 |  | 3 | 13
MiniMental State Exam [Mean (Standard Deviation); unit: units on a scale] — Total score was used. Scores ranged from 0-30. A higher score indicates better cognitive functioning. Population: MMSE data collected on residents only not on staff
  units on a scale
    number analyzed (Participants) | 10 | 0 | 0 | 10
    (all) | 18.8 (3.8) |  |  | 18.8 (3.8)

OUTCOME MEASURES:

1. Primary Outcome: Caregiver Activity Survey
Description: Validated scale requires caregivers to report on amount of time spent caregiving for a particular patient. It has high test-retest reliability. Caregivers will be asked to complete this instrument once every two weeks. The scale describes the total number of minutes spent daily on six different caregiving activities. Therefore the minimum value for each item is 0 and the maximum is 1,440 for each item. Higher scores on each item mean more time spent caregiving.
Time Frame: week 2
Population: TIme reported by professional care giver spent in caring for monitored resident
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Residents in Memory Care or Skilled Nursing Facility | Resident in Independent Living Setting | Care Partners
Number analyzed (Participants) | 0 | 0 | 2
minutes |  |  | 305.7 (177.5)

2. Secondary Outcome: Zarit Caregiver Burden Scale
Description: This is validated instrument designed to reflect what people sometimes feel when taking care of another person. Caregivers will be asked to complete this instrument once every two weeks. Total score was calculated. Scores ranged from 0-48 with a higher score indicating greater caregiver burden.
Time Frame: Up to 6 months
Population: No data were collected for this measure because the nurse practitioners failed to respond to the surveys biweekly.
Arm/Group | Residents in Memory Care or Skilled Nursing Facility | Resident in Independent Living Setting | Care Partners
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: AD Quality of Life Scale
Description: Assesses Caregiver quality of life with 13 questions rating from poor to excellent. Caregivers circle their responses. Caregivers will be asked to complete this instrument once every two weeks. Total score was calculated. Scores ranged from 13-52, with a higher score indicating better quality of life in caregivers.
Time Frame: up to 6 months
Population: No data were collected for this measure because nurse practitioners failed to complete the biweekly survey.
Arm/Group | Residents in Memory Care or Skilled Nursing Facility | Resident in Independent Living Setting | Care Partners
Number analyzed (Participants) | 0 | 0 | 0

4. Other Pre Specified Outcome: Device Accuracy
Description: Percentage of physical checks where device displayed correct location of patient/resident. Only partners reported on the accuracy. No data were required from participants. Therefore, they were entered as 0s in the chart.
Time Frame: First month of overall study period
Population: In validation phase of study, Nursing assistants were sent intermittent prompts to compare location of resident as indicated by the device to actual physical location of patient as determined by direct observation.
Measure: Number; unit: percentage of observations
Units Other Than Participants: observations
Groups:
- Nurse Assistants Recorded Data From Residents in Memory Care or Skilled Nursing Facility: Activlink insole: Dementia patients will wear the provided insole inserted into their own shoes. The insole will have a small electronic sensor that measures acceleration, foot force, and/or orientation.
  Nurse assistants, which are the partner group in the study, reported accuracy of device for each participant. Participants were not required to complete this outcome.
- Partner Reported Data on Resident in Independent Living Setting: Activlink insole: Dementia patients will wear the provided insole inserted into their own shoes. The insole will have a small electronic sensor that measures acceleration, foot force, and/or orientation.
- Residents in Memory Care or Skilled Nursing Facility: residents were not required to report on this outcome
- Resident in Independent Living Setting: participants were not required to report on this outcome
Arm/Group | Nurse Assistants Recorded Data From Residents in Memory Care or Skilled Nursing Facility | Partner Reported Data on Resident in Independent Living Setting | Residents in Memory Care or Skilled Nursing Facility | Resident in Independent Living Setting
Number analyzed (Participants) | 9 | 0 | 0 | 0
Number analyzed (observations) | 9 | 0 | 0 | 0
percentage of observations | 87.83 |  |  |

ADVERSE EVENTS:
Time Frame: Full study period of 6 months for each participant.
Description: Care partners engaged only in observation and survey reporting and were not considered at risk for adverse events of any type including all-cause mortality.
Arm/Group | Residents in Memory Care or Skilled Nursing Facility | Resident in Independent Living Setting | Care Partners
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/0 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/0 | 0/3
Other Adverse Events (participants affected / at risk) | 1/10 | 0/0 | 0/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Residents in Memory Care or Skilled Nursing Facility (N=10) | Resident in Independent Living Setting (N=0) | Care Partners (N=3)
Accurate WiFi-Based Localization of Dementia Patients For Caregiver Support (Product Issues) | 1 (1) | 0 | 0 — Discomfort with fit of product

LIMITATIONS AND CAVEATS:
Participants from study 2A discontinued before the end of the intervention period, and caregiving nurse practitioners failed to respond to the surveys biweekly. Only 4 surveys were collected by the end of study 2A. Largely because of the Corona Virus 19 pandemic all contacted participants from study 2B declined or withdrew consent of baseline data collection and treatment implementation. Therefore, no data were collected for this phase of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-11-02): https://cdn.clinicaltrials.gov/large-docs/19/NCT03360019/Prot_SAP_000.pdf
  • Informed Consent Form (2021-10-06): https://cdn.clinicaltrials.gov/large-docs/19/NCT03360019/ICF_001.pdf